CLINICAL TRIAL: NCT00275314
Title: WP16302 A Bioequivalence Study Comparing Ganciclovir From the Valganciclovir Syrup Formulation and the Commercial Valganciclovir 450mg Tablet (Valcyte®) at a Dose of 900mg in Kidney Transplant Recipients, Sponsor Protocol Dated 8/11/2005 and Investigator Brochure Version August 2005
Brief Title: WP16302 A Bioequivalence Study Comparing Ganciclovir From the Valganciclovir Syrup Formulation and the Commercial Valganciclovir 450mg Tablet (Valcyte®) at a Dose of 900mg in Kidney Transplant Recipients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study never started at our site Funding issue
Sponsor: University of Pittsburgh (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 0512007
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Kidney Transplant
Keywords: transplantation
MeSH Terms: interventions — Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir

SUMMARY:
This is a multi-center, open label, randomized, 3-way cross-over study. 21 subjects will be randomized to receive all three treatments in one of three treatment sequences.

Patients at risk of CMV disease (D+R-, D+R+, D-R+), who are being treated prophylactically with Valcyte® (commercially available tablets), after their first or second kidney transplant and who have adequate renal and hematological function will be eligible for the study. Screening may be at any time after transplantation provided that follow-up procedures can be completed during the scheduled time of prophylaxis. The first dose of study drug may be between 1 and 14 days after screening provided the transplant has stabilized, stable serum creatinine and steady-state kinetics of ganciclovir and calcineurin inhibitor therapy have been attained. Follow-up will take place 7- 14 days after last dose of study drug administration; therefore the duration of the study will be up to 5 weeks.

DETAILED DESCRIPTION:
Each patient will receive 900 mg of Valcyte® daily with food for the period specified in that center (typically 100 days), starting as soon as possible after the transplant. According to routine practice, intravenous ganciclovir (5 mg/kg) may be substituted if the patient is unable to tolerate oral medication, during which time the patient will not be enrolled into the study. The dose of Valganciclovir may be reduced or interrupted at the discretion of the Investigator if he, or she, suspects that ganciclovir-related toxicity has occurred, or if the estimated creatinine clearance of the patient drops below 60 ml/min For the actual study, each patient will receive 2 days treatment on consecutive days with each Valganciclovir syrup formulation (900 mg once a day.) and the tablet formulation (900 mg once a day) in a randomized order, before continuing with Valcyte® prophylaxis (commercially available tablets). The following three treatments will be administered in this study: Randomization will occur through the IDS pharmacy and a computerized system will randomize the subjects.

Treatment A (Reference): Valganciclovir tablets 2 x 450 mg once a day for 2 days

Treatment B (Test): Valganciclovir tutti-frutti flavored syrup, 900 mg once a day for 2 days

Treatment C: (First formulation) Valganciclovir strawberry flavored syrup, 900 mg once a day for 2 days

All formulations will be administered orally within 15 minutes of completion of a standard breakfast (400-800 kcal). Patients will be seen at that GCRC (General Clinic Research Center) on the 8th floor of Montefiore Hospital for all study visits except follow-up. This visit will take place in the Infectious Disease Clinic, 7th floor Falk Clinic.

Screening:

A screening examination will be performed between 1 and 14 days before the start of the study (the day of first dosing with study drug). Patients who fulfill all of the inclusion and none of the exclusion criteria will be accepted on to the study. Patients who fail the renal or hematological function criteria may be re-screened if these parameters improve and if they are still being treated with Valcyte®. The following procedures will be performed to establish each patient's general health and eligibility for enrollment into the study: Record medical history, including etiology of end-stage organ disease, details of transplant (date and type), any previous disease (including CMV) and treatments, immunosuppressive drugs and doses within the previous month or from transplantation, whichever is the shorter, Record CMV serology of donor and recipient., perform physical examination; record demographic information including sex, age and race/ethnicity; Obtain vital signs, height and weight; Draw blood samples for laboratory screening of hematology (about one teaspoon of blood) and routine serum chemistry, including calculation of estimated creatinine clearance; Obtain a mid-stream urine sample for urinalysis and a pregnancy test (females only). This visit will take about 30 minutes. Patient will be seen while in hospital by the research coordinators and research physicians, while recovering from the kidney transplant procedure.

Day 1

Patients will come to the GCRC the evening before, or during the morning of Day 1, within 14 days of screening. The following procedures will be carried out on all patients:

* Assessment that the patient is on stable calcineurin inhibitors and Valganciclovir therapy ( ≥ 4 days); assignment of patient identification number; physical examination; concomitant medication since the last visit will be collected; vital signs and weight; blood samples for hematology and serum chemistry (5 cc); mid-stream sample of urine for urinalysis and pregnancy testing (females of childbearing potential only); and breakfast.
* Study drug will be administered (either two Valganciclovir tablets or 900 mg (18 mL) of syrup formulation of Valganciclovir) with breakfast (must be within 15 minutes of completion of breakfast). Adverse events and concomitant medications will be recorded. Patients may be discharged after dosing. This visit will take about 2-3 hours to complete.

Days 2, 4 and 6

Patients will return to the GCRC during the morning of these days. The following procedures will be carried out on all patients:

* Pre-dose PK blood sample for determination of trough levels of ganciclovir (5cc)
* Breakfast will start within 15 minutes of the pre-dose PK blood sample. The study drug (either two Valganciclovir tablets or 900 mg (18 mL) of syrup formulation of Valganciclovir) will be administered with breakfast (must be within 15 minutes of completion of breakfast).
* The following procedures will be carried out after dosing: pharmacokinetic blood samples (total blood collected each day is 11cc) for determination of plasma levels of ganciclovir 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0, and 12 hours post-dose (time windows of ± 5 minutes are allowed for all samples up to 4 hours and ± 20 minutes for samples between 6 and 12 hours)
* Adverse events and concomitant medications will be documented. Patients may be discharged after the 12-hour sample. This day will take twelve -thirteen hours to complete.

Days 3 and 5

Patients will return to the GCRC during the morning. The following procedures will be carried out on all patients:

* Vital signs and weight; 24 hour PK blood sample (± 30 minutes) for determination of trough levels of ganciclovir before dosing with the next formulation of study drug (1cc); Breakfast will start within 15 minutes of the pre-dose PK blood sample.
* Study drug will be administer (either two Valganciclovir tablets or 900 mg (18 mL) of syrup formulation of Valganciclovir) with breakfast (must be within 15 minutes of completion of breakfast). Adverse events and concomitant medications will be recorded. Patients may be discharged after dosing. This visit will take about 2-3 hours to complete.

Day 7

Patients will return to the GCRC during the morning. The following procedures will be carried out on all patients:

* Blood samples for hematology and serum chemistry (5cc); mid-stream sample of urine for urinalysis; 24 hour PK blood sample (± 30 minutes) for determination of trough levels of ganciclovir before dosing (5cc). Breakfast will start within 15 minutes of the pre-dose PK blood sample.
* Two Valcyte® tablets will be administered (supplied by the center) with breakfast (must be within 15 minutes of completion of breakfast). Adverse events and concomitant medications will be recorded and patients may then be discharged from the GCRC. This visit will take about 2-3 hours to complete.

During the Study The following safety assessments will be made throughout the study, from screening to follow-up, as applicable: adverse events (AE's), including rejection and graft loss, opportunistic infections (CMV and others) and treatments; concomitant treatments, including immunosuppressive therapy (induction, maintenance and treatment of rejection) and patient survival will be documented.

Follow-up Phase Patients will return between Days 13 to 20 for follow-up. The follow-up procedures will include a physical examination, body weight, vital signs, clinical laboratory safety tests (hematology, serum chemistry and urinalysis) (5cc), urine pregnancy test (females of childbearing potential only) and the recording of adverse events and concomitant medications. Once this visit is complete the patient will have completed the study. This visit should take about one hour to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has received first or second kidney transplant.
2. Transplantation occurred at least 14 days before screening.
3. Patient at risk of CMV disease (serostatus, D+R-, D+R+ or D-R+).
4. Patient aged 18 to 68 years inclusive.
5. Patient able to tolerate oral medication from screening to follow-up.
6. Patient being treated with Valganciclovir for prophylaxis of CMV disease according to current center practice.
7. Patient on stable calcineurin inhibitor and 900 mg Valganciclovir therapy (≥ 4 days prior to Day 1).
8. Patient with stable serum creatinine (± 0.2 mg/dL) for duration of at least 4 days prior to dosing on Day 1.
9. Patient with adequate hematological and renal function defined as:

   * Estimated creatinine clearance ≥ 60 ml/min
   * Absolute neutrophil count ≥ 2500 cells/µL
   * Platelet count ≥ 100,000 cells/µL
   * Hemoglobin ≥ 9.0g/dL
10. Patient agrees to use an effective method of contraception (or abstinence from sexual activity) throughout the study period and for 90 days after follow-up, if female of child-bearing potential, or if male with a female partner of child-bearing potential.
11. Females of childbearing potential with a negative pregnancy test at screening.
12. Patient able to participate, willing to give written, informed consent and comply with the study restrictions.

    -

Exclusion Criteria:

* Patients with any of the following will be excluded from the study:

  1. Patient is simultaneously participating in another clinical trial, except as approved by the Sponsor.
  2. Patient has used an investigational drug within three months of screening.
  3. Patient has exhibited in the past an allergic, or other significant adverse reaction to acyclovir, Val acyclovir, ganciclovir or Valganciclovir.
  4. Patient has severe, uncontrolled diarrhea.
  5. Evidence of graft rejection as determined by the Investigator.
  6. Patient requires the use of any prohibited concomitant medications (Section 4.4).
  7. Patient has previously participated (i.e. completed Day 1) in this clinical trial.
  8. Patient is pregnant or a lactating female who will not discontinue nursing prior to study entry.
  9. Patient has received anti-CMV prophylaxis with a treatment other than intravenous cytogam, intravenous ganciclovir or Valganciclovir between transplant and enrollment.
  10. Patient with active bacterial, viral, fungal or protozoal infection.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5
Dates: Start 2006-02; Study Completion 2006-04

PRIMARY OUTCOMES:
The primary objective of the study is to determine bioequivalence of ganciclovir from the
Valganciclovir tutti-frutti syrup formulation and the 450 mg tablet formulation at a dose of 900 mg administered in the fed state.

SECONDARY OUTCOMES:
The secondary objective is to compare the systemic exposure to ganciclovir from the
Valganciclovir strawberry syrup formulation with the valganciclovir tutti-frutti syrup formulation at a dose of 900mg.

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States